CLINICAL TRIAL: NCT04047355
Title: A Pilot/Feasibility Study of the Use of High Dose Propranolol to Treat Severe and Chronic Challenging Behaviors in Adolescents and Adults With Autism Spectrum Disorders
Brief Title: Propranolol for Challenging Behaviors in Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: New Jersey Governor's Council for Medical Research and Treatment of Autism (Unknown); New York State Institute for Basic Research (Other Government)
Responsible Party: Principal Investigator, Barbie Zimmerman-Bier, M.D., Assistant Professor of Pediatrics, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro20170001942; CAUT17 APL025 (Other Grant/Funding Number: NJ Governor's Council)
Record Dates: First submitted 2019-07-12; First posted 2019-08-06 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder; Developmental Disability; Aggression; Self-Injurious Behavior; Challenging Behavior
Keywords: Propranolol; Beta Blocker; Psychopharmacology; Inderal
MeSH Terms: conditions — Autism Spectrum Disorder; Developmental Disabilities; Aggression; Self-Injurious Behavior | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Propranolol first (Experimental): Participants randomly assigned to this group will receive Propranolol first. After the washout period, they will receive Placebo.
  Propranolol will be given in liquid or pill form.
  Interventions: Drug: Propranolol
- Group B: Placebo first (Placebo Comparator): Participants randomly assigned to this group will receive Placebo first. After the washout period, they will receive Propranolol.
  Placebo will look identical to the study drug Propranolol.
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — Propranolol is a beta-blocker used to treat high blood pressure, irregular heartbeats, and tremors. It is used after a heart attack and to prevent migraine headaches and chest pain. It is also used off-label for anxiety and PTSD.
  Other Names: Inderal

SUMMARY:
Severe challenging behaviors such as aggression and self-injury can cause significant morbidity and decrease the quality of life for individuals with Autism Spectrum Disorders (ASD). There are only two medications (Risperdal and Abilify) rigorously studied and FDA-approved for the treatment of irritability in individuals with ASD. These medications are not always successful and have many short and long-term side effects. Well-designed studies demonstrating efficacy and safety of alternative medication treatment choices are needed. There is preliminary evidence that high-dose propranolol can be effective in individuals with ASD who display severe aggression and have not responded to antipsychotics or mood stabilizers. Concerns regarding the safety of high dose propranolol have limited its clinical application. Well-designed clinical trials demonstrating the efficacy and safety of high dose propranolol will have significant effects on clinical practice and improve the physical and behavioral quality of life for an underserved subset of individuals with ASD.

This study will pilot the safety and efficacy of high dose propranolol. The investigators will randomly assign participants to either propranolol or to placebo later crossing each participant over to the other group. As propranolol can cause changes in blood pressure and heart function, each participant will complete initial comprehensive testing to monitor cardiac safety throughout the study. The investigators will be utilizing telemedicine and computer based telemetry to minimize the burden of office visits on the individual and family.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo controlled crossover study. A complete cardiac exam will be conducted by the pediatric cardiology team at the Robert Wood Johnson Medical School. All participants will remain on their existing, pre-study medication throughout all phases of the study.

Once admitted to the study, a baseline period will begin. During the baseline period, cognitive and adaptive information will be collected. The participant will then be randomly assigned to propranolol (Phase A) or placebo (Phase B). The titration schedule will be flexible and the dose can be held steady for an extended period. Dose reduction to manage side effects are allowed at any time. Each week the family will complete behavioral forms online and meet with the study psychiatrist via telemedicine. Following the initial Phase (A or B), participants will undergo a washout period (whether propranolol or placebo). Then, they will crossover to the other Phase (A or B). Upon completion of the crossover phase, the study blind will be broken. The participants then had the option of enrolling in an open label study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 12-30 years and is a resident in the state of New Jersey.
2. Diagnosis of autism conducted by a clinician with confirmation using the Autism Diagnostic Observation Schedule (ADOS) or the Social Communication Questionnaire (SCQ).
3. At least one of the following challenging behaviors.

   1. Self-injurious behaviors (e.g., hitting one's self, head banging or banging of other body parts causing some degree of tissue damage);
   2. Physical aggression towards others (e.g., hitting, kicking, pushing, or throwing objects at others);
   3. Disruptive behaviors including property destruction during anger episodes, excessive screaming which interferes with functioning; and
   4. The challenging behaviors are generally (but not necessarily exclusively) associated with a congruent affect (i.e. anger or rage when aggressing) as determined by the study psychiatrist.
4. Pharmacologic treatment with at least two psychotropic including one antipsychotic medication has yielded inadequate outcome (partial improvement on one or more medications is acceptable for the study).
5. Clinical Global Impression Severity scale score of 6 or 7.
6. Aberrant Behavior Checklist--Community Irritability scale score at or above 18.
7. Medical and cardiac clearance.

Exclusion Criteria:

1. Asthma or any history of asthma or any disorder involving bronchoconstriction.
2. Cardiac Diseases in which the use of propranolol at high doses would be contraindicated.
3. Uncontrolled Seizure disorder (participant had a seizure within the past year and/or changes in seizure medication in the previous six months).
4. Diabetes or a history of ketoacidosis.
5. Any other medical disorder or medication which would contraindicate the use of propranolol.
6. History of allergy or adverse reaction to propranolol.
7. Pregnancy.
8. Medication exclusions include clonidine/guanfacine / digoxin or other medications affecting blood pressure.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbie Zimmerman-Bier, M.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Department of Pediatrics, Division of Pediatric Neurology, Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a crossover study. 6 subjects underwent both experimental phases (i.e., crossover design). 3 subjects underwent Propranolol first, then Placebo while the remaining 3 subjects underwent Placebo first, then Propranolol.
Groups:
- Group A: Propranolol First, Then Placebo Second: First Propranolol, then Placebo, then Open Label Propranolol.
  Participants randomly assigned to this group received Propranolol first. Titration time period and maximum dose were flexible based on individual response. Maximum dose was up to 200 mg TID for 6 weeks.
  After the washout period, they received Placebo in the same fashion.
- Group B: Placebo First, Then Propranolol Second: First Placebo, then Propranolol, then Open Label Propranolol.
  Participants randomly assigned to this group received Placebo first. After the washout period, they received Propranolol. Titration time period and maximum dose were flexible based on individual response. Maximum dose was up to 200 mg TID for 6 weeks.
Period: Overall Study
Arm/Group | Group A: Propranolol First, Then Placebo Second | Group B: Placebo First, Then Propranolol Second
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants underwent baseline phase. The primary measure during baseline and all phases thereafter was the Aberrant Behavior Checklist--Community Irritability Subscale.
Groups:
- Group A: First Propranolol, Then Placebo: Participants randomly assigned to this group received Propranolol first. After the washout period, they received Placebo.
- Group B: First Placebo, Then Propranolol: Participants randomly assigned to this group received Placebo first. After the washout period, they received Propranolol.
- Total: Total of all reporting groups
Arm/Group | Group A: First Propranolol, Then Placebo | Group B: First Placebo, Then Propranolol | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Full Range); unit: years] | 15 [13 to 19] | 15 [13 to 18] | 15 [13 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Aberrant Behavior Checklist--Community (ABC-C) Irritability Subscale Scores
Description: The Aberrant Behavior Checklist--Community (ABC-C) is a behavior checklist that measures drug and other treatment effects in people with intellectual and developmental disabilities. It is made up of five subscales, including Irritability, Lethargy, Inappropriate Speech, Hyperactivity, and Stereotypy based on 58 items that describe various behavioral problems. Each item is scored on a Likert scale: 1 = not at all a problem, to 3 = problem is severe in degree. The Irritability Subscale served as the primary dependent measure. The minimum score on the Irritability Subscale is 0 and the maximum score is 45. Lower scores represent better outcome.
Time Frame: Titration schedule varied based on individual response; it was not predetermined. On average, Placebo was 8 wks and Propranolol was 11 wks, including titration. The last Baseline score and the last scores from Placebo and Propranolol phases were analyzed.
Population: Participants served as their own controls. Each participant received both Propranolol and Placebo. The treatment order was randomized.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Propranolol Phase: All 6 participants received propranolol either as the first treatment or the second treatment.
- Placebo Phase: All 6 participants received placebo either as the first treatment or the second treatment.
Arm/Group | Propranolol Phase | Placebo Phase
Number analyzed (Participants) | 6 | 6
score on a scale | 14.0 [6.25 to 16.50] | 18.50 [12.25 to 27.25]
Statistical Analysis 1: Comparison: Propranolol Phase vs Placebo Phase; A post-hoc power analysis was conducted using G*Power, v. 3.1, to determine the achieved power for the Wilcoxon signed-rank test for matched pairs; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney) — The a-priori threshold for statistical significance was set at α = 0.05; Median Difference (Final Values) = 3.00 — The placebo phase serves as the control condition and the propranolol phase serves as the treatment condition
Statistical Analysis 2: Comparison: Propranolol Phase vs Placebo Phase; Test type: Superiority; Effect size (r) = -0.64
Statistical Analysis 3: Comparison: Propranolol Phase vs Placebo Phase; Test type: Superiority; Post-hoc power analysis = 0.39 — The alpha error probability was set at α = 0.05 (two-tailed)

2. Secondary Outcome: Clinical Global Impression Improvement (CGI-I) Scale
Description: The Clinical Global Impression Improvement (CGI-I) scale is used by the study psychiatrist to judge the overall clinical condition relative to baseline using the same scale as the CGI-S. The study psychiatrist will rate the improvement from baseline. The CGI consists of a 7-point subjective scale assessing symptom. Lower scores represent better outcomes. Scores of 1, 2, and 3 represent normal, some presence of symptoms, and mild behavior, respectively. A score of 4 represents moderate behavior. Scores of 5, 6, and 7 represent marked, severe, and among the most severe behavior, respectively.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Propranolol Phase; Placebo Phase: All participants received propranolol either as the first treatment or the second treatment.
Arm/Group | Propranolol Phase | Placebo Phase
Number analyzed (Participants) | 6 | 6
score on a scale | 2.00 [1.75 to 3.50] | 5.50 [3.75 to 6.00]
Statistical Analysis 1: Comparison: Propranolol Phase vs Placebo Phase; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney) — The a-priori threshold for statistical significance was set at α = 0.05; Median Difference (Final Values) = 2.00 — The placebo phase serves as the control condition and the propranolol phase serves as the treatment condition
Statistical Analysis 2: Comparison: Propranolol Phase vs Placebo Phase; Test type: Superiority; Effect size (r) = -0.74
Statistical Analysis 3: Comparison: Propranolol Phase vs Placebo Phase; Test type: Superiority; Post-hoc power analysis = 0.59 — The alpha error probability was set at α = 0.05 (two-tailed)

ADVERSE EVENTS:
Time Frame: Weekly over the entire double-blind portion of the study. Exact duration varied per participant due to individualized titration periods (approximately 5-7 months based on individual titration schedule). The open label phase was two months.
Groups:
- Propranolol: Subjects who received Blinded Propranolol
- Placebo: Subjects who received Placebo
- Open Label: Subjects who received Open Label Propranolol
Arm/Group | Propranolol | Placebo | Open Label
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 2/6 | 0/6 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol (N=6) | Placebo (N=6) | Open Label (N=5)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT04047355/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT04047355/ICF_001.pdf